CLINICAL TRIAL: NCT05502952
Title: Combined Microneedling and Topical Pentoxifylline Vesrus Intalesional Pentoxifylline in Treatment of Alopecia Areata: Intra-indiviual Comparative Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Manar Ibrahim Abdelhameed, assistent lecturer at dermatology,venerology and andrology department, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-22-07-24
Record Dates: First submitted 2022-07-26; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — Pentoxifylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alopecia areata (Experimental)
  Interventions: Drug: Pentoxifylline

INTERVENTIONS:
Drug: Pentoxifylline — Combined microneedling and topicalpentoxifylline vesrus intalesional pentoxifylline in Alopecia Areata patches in the same patient

SUMMARY:
Alopecia areata (AA) is a common autoimmune disease that targets hair follicles with a prevalence of approximately 0.1% and a lifetime incidence of approximately 1.7%. AA is the third most prevalent nonscarring hair loss disease. Pentoxifylline (PTX) is a non-selective inhibitor of phosphodiesterases, which moderates the intracellular levels of cyclic adenosine monophosphate and cyclic guanosine monophosphate by decreasing their hydrolysis and augmenting cyclic nucleotide-dependent signal transduction which leads to a wide spectrum of effects on the inflammation. PTX has anti inflammatory effects by inhibiting the pro-inflammatory cytokines (eg, IL-1, IL-6, and IL-8).Intralesional therapy has a number of advantages over topical therapy, including a faster and longer duration of action, penetration that is deeper than topical therapy, removal of the need for long-term topical medication, and improved patient compliance.The effect of microneedling for treatment of AA is supposed to stimulate the dermal papilla and stem cells by mechanical trauma and increasing the blood supply to the hair follicles.

ELIGIBILITY:
Inclusion Criteria:

* All patients over the age of 18 years of both sex, with a clinical diagnosis of localised AA of two or more AA scalp patches in the same patient.

Exclusion Criteria:

* Patients who received systemic or topical treatment for A.A in the previous three months prior to the start of the study.
* Patients who are pregnant or lactating.
* Patients who have bleeding or coagulation disorders.
* Patients with autoimmune diseases, liver, or renal diseases were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
measuerement of improvement of alopecia areata patches by SALT score | 12 month
  The clinical response will be evaluated based on the SALT score, the following percentages of scalp hair regrowth are possible: A0 = no change or further loss, A1 = 1%-24% regrowth, A2 = 25%-49% regrowth, A3 = 50%-74% regrowth, A4 = 75%-99% regrowth, and A5 = 100% regrowth.
measuerement of improvement of alopecia areata patches by Trichoscopic signs | 12 month
  Trichoscopic examination each visit to evaluate the results and record signs of improvement of the disease including (short vellus hairs and terminal hairs) and disappearance of signs of activity(exclamation marks, blackdots)

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] El Taieb MA, Hegazy EM, Ibrahim HM, Osman AB, Abualhamd M. Topical calcipotriol vs narrowband ultraviolet B in treatment of alopecia areata: a randomized-controlled trial. Arch Dermatol Res. 2019 Oct;311(8):629-636. doi: 10.1007/s00403-019-01943-8. Epub 2019 Jun 24. PMID 31236672
- [Background] Lai VWY, Chen G, Gin D, Sinclair R. Cyclosporine for moderate-to-severe alopecia areata: A double-blind, randomized, placebo-controlled clinical trial of efficacy and safety. J Am Acad Dermatol. 2019 Sep;81(3):694-701. doi: 10.1016/j.jaad.2019.04.053. Epub 2019 Apr 30. PMID 31048013
- [Background] El-Taweel AI, Akl EM. Intralesional pentoxifylline injection in localized alopecia areata. J Cosmet Dermatol. 2019 Apr;18(2):602-607. doi: 10.1111/jocd.12796. Epub 2018 Oct 9. PMID 30302901
- [Background] Fukumoto T, Fukumoto R, Magno E, Oka M, Nishigori C, Horita N. Treatments for alopecia areata: A systematic review and network meta-analysis. Dermatol Ther. 2021 May;34(3):e14916. doi: 10.1111/dth.14916. Epub 2021 Mar 4. PMID 33631058